CLINICAL TRIAL: NCT05703737
Title: Respiratory Function and Respiratory Muscle Strength in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Collaborators: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: karanki2
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; pulmonary function; respiratory muscle strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, which aims to evaluate the respiratory functions and respiratory muscle strength of individuals with Adolescent Idiopathic Scoliosis (AIS), it is planned to investigate the relationship between the respiratory parameters obtained and the severity, type, location of the curvature, rotation angle and wearing brace.

The population of the study consists of individuals with AIS, and the sample consists of individuals with AIS followed in the Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Orthopedics and Traumatology Clinic. For this purpose, it was planned to include at least 60 individuals with AIS, aged 10 years and older, with at least 20 degrees of scoliotic curvature, who applied to the clinic for the first time or came for control.

Pulmonary Function Tests (PFT) will be applied to evaluate the respiratory functions of the participants involved, and intraoral pressure measurement (MIP, MEP) will be applied to evaluate the inspiratory and expiratory muscle strengths; The severity of the scoliotic curvature will be measured with the Cobb method on the same day's radiograph, and the axial rotation angle will be measured with the Scoliometer.

IBM Statistical Package for Social Sciences Version 24 statistical program will be used in the analysis of the data. Continuous variables will be given as mean ± standard deviation, qualitative variables as numbers and percentages.

Pearson Correlation analysis will be used for the relationship between the variables, Independent Samples t-test will be used for the comparison of independent groups, and statistical significance will be taken as p≤0.05 in all measurements.

It is thought that this planned study will contribute to studies evaluating the respiratory functions and respiratory muscle strength of individuals with AIS, which have been designed in different types and reported different results in the literature.

Evidence-based data obtained by determining the clinical parameters associated with these values are expected to guide clinicians in terms of being holistic in the treatment of individuals with scoliosis, and in which situations and for what purpose pulmonary rehabilitation approaches should be included.

DETAILED DESCRIPTION:
Scoliosis is a complex three-dimensional deformity characterized by a lateral deviation of the spine of at least 10 degrees in the coronal plane. Scoliosis, which develops due to many reasons, is called "Adolescent Idiopathic Scoliosis (AIS)" if it occurs in the period from the onset of puberty to the closure of the growth plates.

The main treatment options for scoliosis are; Known as observation, orthosis and surgical intervention, the choice of the most appropriate treatment depends on the patient's age, menarche status, location and size of the curvature, and risk of progression.

Scoliosis can cause a significant increase in respiratory workload by directly decreasing chest wall compliance and indirectly reducing lung compliance. Abnormal ventilation patterns, especially restrictive ventilatory disorders, are seen in individuals with AIS, especially in curves greater than 45°; Sagittal diameter of the thorax, total lung area and especially vertebral rotation at T8-T9 levels can affect respiratory functions. In a study, it was shown that patients with mild or moderate idiopathic scoliosis had significantly lower Forced Vital Capacity (FVC) values compared to healthy controls. On the other hand, in a recent study in which 30 individuals with scoliosis were included, FVC values were found to be low in only two cases, which was thought to be due to the fact that the curve intensities of the participants were mild (Cobb angle< 20ᴼ). In the literature, studies examining the relationship between location, type, angle of rotation, presence of brace and duration of use, apart from the severity of the curvature, and pulmonary functions in individuals with AIS are insufficient. Low FEV1 and FVC values were found in 19% of AIS patients who had pulmonary function test preoperatively, and individuals with high grade (Cobb angle > 70ᴼ) and wide main thoracic type curves were reported to be more affected. Although no significant results were obtained in the degree of axial rotation in the same study, it was observed that the rotation angles of the cases with low PFT parameters were higher. A different study reported that the size of the thoracic curve and the number of involved vertebrae were negatively correlated with pulmonary parameters in individuals with AIS, and that spirometric examination is necessary, especially in surgical planning. Although studies have shown that respiratory muscle strength of individuals with AIS is decreased compared to healthy controls, even with mild curvatures, the cause of muscle dysfunction is not known exactly and it is thought that several factors may affect muscle function (nutritional status, physical activity, systemic inflammation, etc.). In scoliosis, especially the distortion of the thorax, the placement of the diaphragm and intercostal muscles and affecting the force production can also reduce respiratory muscle strength. In a study, a weak correlation was found between the angular value of scoliosis and respiratory muscle strength in individuals with AIS, and it was reported that respiratory muscle strength may be associated with physical deconditioning. In individuals with a high progression rate and an indication for scoliosis surgery, decreased respiratory muscle strength before surgery may cause a serious increase in respiratory workload, causing the patient to be unable to extubat, and post-operative respiratory failure due to respiratory muscle weakness. Therefore, respiratory muscle strength and function levels are important in curves with a high progression rate and surgery is planned, and it is important to use methods that prevent and reduce respiratory muscle dysfunction.

In the literature, studies evaluating respiratory muscle strength and related parameters of individuals with AIS are very limited. In our study, it was aimed to measure the respiratory functions and respiratory muscle strength of individuals with AIS objectively and to investigate the relationship of these values with the severity of curvature, type, location, rotation angle and corset use. It is expected that the evidence-based data obtained will guide the treatment of individuals with scoliosis to be holistic and in which situations and for what purpose pulmonary rehabilitation approaches should be included.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* 10 years and older
* Having been diagnosed with Adolescent Idiopathic Scoliosis,
* At least 20 degrees of scoliotic curvature in the coronal plane

Exclusion Criteria:

* Individuals aged 9 and under, 20 years and over
* Individuals with neuromuscular and congenital scoliosis
* Individuals with pulmonary dysfunction due to a different pathology
* Individuals with a history of surgery
* Cases with mental retardation
* Individuals who do not understand, cannot apply, and cannot cooperate with respiratory tests

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases with Adolescent Idiopathic Scoliosis followed in a Prof. Dr. Suleyman Yalcin City Hospital (Secondary health institution)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
FEV1 (liter) | During the 3-month data collection process, pulmonary function measurements are made on the same day as the day the participants came to the hospital for examination or control.
  This is the amount of air with pulmonary function test that the patient can force out of their lungs in one second.
FEV1 (%-percentage) | During the 3-month data collection process, pulmonary function measurements are made on the same day as the day the participants came to the hospital for examination or control.
  This is the percentage of air with pulmonary function test that the patient can force out of their lungs in one second.
FVC (liter) | During the 3-month data collection process, pulmonary function measurements are made on the same day as the day the participants came to the hospital for examination or control.
  This is the greatest total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FVC (%-percentage) | During the 3-month data collection process, pulmonary function measurements are made on the same day as the day the participants came to the hospital for examination or control.
  This is the percentage of total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FEV1/FVC (percentage) | During the 3-month data collection process, pulmonary function measurements are made on the same day as the day the participants came to the hospital for examination or control.
  The FEV1/FVC ratio is a number that represents the percentage of patient lung capacity patient is able to exhale in one second.
Inspiratory muscle test | During the 3-month data collection process, intraoral pressure measurements are made on the same day as the day the participants came to the hospital for examination or control.
  Maximal inspiratory pressure (MIP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Expiratory muscle test | During the 3-month data collection process, intraoral pressure measurements are made on the same day as the day the participants came to the hospital for examination or control.
  Maximal expiratory pressure (MEP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).

SECONDARY OUTCOMES:
Cobb method | During the 3-month data collection process, Cobb measurements are made on the same day as the day the participants came to the hospital for examination or control.
  It is the standard measurement method used in coronal grading of the angle of scoliotic curvature on anteroposterior radiography. On the graph, the angle between the lines drawn parallel to the upper vertebral edge of the curvature at the upper end and the lower edge of the vertebrae at the lower end gives the cobb angle (Morrissy et al, 1990; Pruijs JE et al, 1994). In order to prevent differences between measurements, measurements are made by the same researcher with the same equipment.
Scoliometer | During the 3-month data collection process, axial trunk rotation measurements are made on the same day as the day the participants came to the hospital for examination or control.
  It is a practical, noninvasive, valid and reliable measurement method used in the objective evaluation of axial trunk rotation. During scoliometer measurement, patients lean forward until their torso is parallel to the ground and hold their torso upright with their arms hanging down (Amendt et al, 1990; Coelho et al, 2013). In our study, the maximum trunk axial rotation value in the thoracic and lumbar regions is evaluated by the same investigator with the same Scoliometer (Orthopedic Systems Inc, Hayward, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: İrem Çetinkaya, MSc, Principal Investigator — Haliç University; Tuğba Kuru Çolak, Phd, Study Director — Marmara University; Seda Saka, Phd, Principal Investigator — Haliç University; Mehmet Fatih Korkmaz, Phd, Study Chair — İstanbul Medeniyet University
Locations (1):
- Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Amaricai E, Suciu O, Onofrei RR, Miclaus RS, Iacob RE, Catan L, Popoiu CM, Cerbu S, Boia E. Respiratory function, functional capacity, and physical activity behaviours in children and adolescents with scoliosis. J Int Med Res. 2020 Apr;48(4):300060519895093. doi: 10.1177/0300060519895093. Epub 2019 Dec 31. PMID 31889450
- [Background] Yildirim S, Ozyilmaz S, Elmadag NM, Yabaci A. Effects of Core Stabilization Exercises on Pulmonary Function, Respiratory Muscle Strength, Peripheral Muscle Strength, Functional Capacity, and Perceived Appearance in Children With Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Aug 1;101(8):719-725. doi: 10.1097/PHM.0000000000001984. Epub 2022 Feb 2. PMID 35859288
- [Background] Johnston CE, Richards BS, Sucato DJ, Bridwell KH, Lenke LG, Erickson M; Spinal Deformity Study Group. Correlation of preoperative deformity magnitude and pulmonary function tests in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2011 Jun 15;36(14):1096-102. doi: 10.1097/BRS.0b013e3181f8c931. PMID 21270699
- [Background] dos Santos Alves VL, Stirbulov R, Avanzi O. Impact of a physical rehabilitation program on the respiratory function of adolescents with idiopathic scoliosis. Chest. 2006 Aug;130(2):500-5. doi: 10.1378/chest.130.2.500. PMID 16899851
- [Background] Koumbourlis AC. Scoliosis and the respiratory system. Paediatr Respir Rev. 2006 Jun;7(2):152-60. doi: 10.1016/j.prrv.2006.04.009. Epub 2006 Jun 2. PMID 16765303
- [Background] Durmala J, Tomalak W, Kotwicki T. Function of the respiratory system in patients with idiopathic scoliosis: reasons for impairment and methods of evaluation. Stud Health Technol Inform. 2008;135:237-45. PMID 18401094
- [Background] Ulubay G, Dilektasli AG, Borekci S, Yildiz O, Kiyan E, Gemicioglu B, Saryal S. Turkish Thoracic Society Consensus Report: Interpretation of Spirometry. Turk Thorac J. 2019 Jan 1;20(1):69-89. doi: 10.5152/TurkThoracJ.2018.180175. PMID 30664428
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Morrissy RT, Goldsmith GS, Hall EC, Kehl D, Cowie GH. Measurement of the Cobb angle on radiographs of patients who have scoliosis. Evaluation of intrinsic error. J Bone Joint Surg Am. 1990 Mar;72(3):320-7. PMID 2312527
- [Background] Pruijs JE, Hageman MA, Keessen W, van der Meer R, van Wieringen JC. Variation in Cobb angle measurements in scoliosis. Skeletal Radiol. 1994 Oct;23(7):517-20. doi: 10.1007/BF00223081. PMID 7824978
- [Background] Amendt LE, Ause-Ellias KL, Eybers JL, Wadsworth CT, Nielsen DH, Weinstein SL. Validity and reliability testing of the Scoliometer. Phys Ther. 1990 Feb;70(2):108-17. doi: 10.1093/ptj/70.2.108. PMID 2296610
- [Background] Coelho DM, Bonagamba GH, Oliveira AS. Scoliometer measurements of patients with idiopathic scoliosis. Braz J Phys Ther. 2013 Mar-Apr;17(2):179-84. doi: 10.1590/S1413-35552012005000081. PMID 23778766